CLINICAL TRIAL: NCT04980690
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability and Efficacy of IBC0966 in Patients With Advanced Malignant Tumors
Brief Title: Clinical Trial of IBC0966 in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IBC0966-I/IIa
Record Dates: First submitted 2021-07-08; First posted 2021-07-28 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Advanced Malignant Tumors
Keywords: PD-L1; CD47; Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Phase Ia - Dose escalation(Acceleration Stage) (Experimental): Phase Ia is an open, non-random, single-arm dose escalation design.
  Acceleration Stage: The initial increasing dose is 0.025 mg/kg, and the dose is increased in 100% increments. Each dose group will enroll 1 subject.
  Interventions: Biological: IBC0966
- Phase Ia - Dose escalation(3+3 Stage) (Experimental): Phase Ia is an open, non-random, single-arm dose escalation design.
  3+3 Stage: The dose is increased in 30%-50% increments between adjacent dose groups, and the increment is determined by the investigator and the sponsor based on the safety data obtained in the previous period.Each dose group will enroll 3 to 6 evaluable subjects (evaluable: at least complete the DLT observation period), and this period continues until the maximum tolerated dose (MTD) is reached.
  Interventions: Biological: IBC0966
- Phase Ib - Dose extension (Experimental): Phase Ib is an open, non-random, single-arm, multi-center research design.
  When phase Ia is transformed into 3+3 stage, a certain dose group meets the conditions for increasing the next dose group (after the DLT observation period of the last subject in the dose group has passed, the safety assessment of the current dose group will be completed) , The dose extension study of this dose group can be carried out, and 6 evaluable (evaluable: at least 2 cycles of dosing and observation) subjects with advanced malignant tumors who have failed standard treatments will be included in this dose group.
  Interventions: Biological: IBC0966
- Phase IIa - Clinical Exploratory Stage(Group A) (Experimental): The Phase IIa is planned to be divided into four indication groups, all of which are open, non-randomized, two-stage, single-arm research design.
  Group A: Recurrent or metastatic triple-negative breast cancer that failed standard treatment.
  Interventions: Biological: IBC0966
- Phase IIa - Clinical Exploratory Stage(Group B) (Experimental): The Phase IIa is planned to be divided into four indication groups, all of which are open, non-randomized, two-stage, single-arm research design.
  Group B: Locally advanced/metastatic non-small cell lung cancer without driver gene mutations that failed standard treatment.
  Interventions: Biological: IBC0966
- Phase IIa - Clinical Exploratory Stage(Group C) (Experimental): The Phase IIa is planned to be divided into four indication groups, all of which are open, non-randomized, two-stage, single-arm research design.
  Group C: Recurrent or metastatic head and neck squamous cell carcinoma that failed standard treatment.
  Interventions: Biological: IBC0966
- Phase IIa - Clinical Exploratory Stage(Group D) (Experimental): The Phase IIa is planned to be divided into four indication groups, all of which are open, non-randomized, two-stage, single-arm research design.
  Group D: Recurrent or metastatic peripheral T-cell lymphoma that failed standard treatment.
  Interventions: Biological: IBC0966

INTERVENTIONS:
Biological: IBC0966 — IBC0966 is an investigational product.

SUMMARY:
This is a phase I/IIa study to evaluate the safety, tolerability and efficacy of IBC0966 for the treatment of subjects with advanced malignant tumors.

DETAILED DESCRIPTION:
The study includes three phases: dose escalation (Phase Ia), dose extension (Phase Ib), and clinical exploration (Phase IIa).

First, the Phase Ia dose escalation will be carried out. After switching to the 3+3 escalation mode, the Phase Ib dose extension study can be carried out at the same time. After Phase Ia is completed and RP2D is obtained, Phase IIa clinical exploratory research can be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old male and female.
2. Phase I (including phase Ia and phase Ib) will enroll patients with advanced malignant tumors who have failed standard treatments.
3. Phase IIa Study-Group A: Recurrent or metastatic triple-negative breast cancer diagnosed by histopathology that has failed standard treatments. Triple-negative breast cancer is defined as estrogen receptor (ER), progesterone receptor (PR), and human epidermis Growth factor receptors (HER2) are all negative.
4. Phase IIa Study-Group B: Advanced/metastatic non-small cell lung cancer with no driver gene mutations that has failed standard treatment confirmed by histopathology.
5. Phase IIa Study-Group C: Recurrent or metastatic head and neck squamous cell carcinoma that failed standard treatments confirmed by histopathology: including nasopharyngeal carcinoma and non-nasopharyngeal head and neck squamous cell carcinoma.
6. Phase IIa study-Group D: Recurrent or metastatic peripheral T-cell lymphoma (PTCL) diagnosed by histopathology that failed standard treatment: Including non-specific PTCL, NK/T-cell lymphoma (nasal type), and angioimmunoblast Cellular T cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL), subcutaneous panniculitis-like T cell lymphoma, enteropathic T cell lymphoma (EATL), and hepatosplenic T cell lymphoma (HSTL) Wait.
7. According to RECIST 1.1 or Lugano 2014 standards, there is at least one measurable lesion, and the measurable lesion has not received local treatment (including local radiotherapy, ablation, and interventional therapy).
8. Agree to provide previously stored tumor tissue specimens or perform a biopsy to collect tumor lesion tissue and send it to the central laboratory for PD-L1 expression level detection and TMB detection.
9. ECOG performance status 0-2.
10. Laboratory examination should meet: ① Blood routine: hemoglobin (HGB) ≥100 g/L, white blood cell count (WBC) ≥3.0×10^9/L, neutrophil count (ANC) ≥1.5×10^9/L, platelet count ( PLT) ≥75×10^9/L; ②Blood biochemistry: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN, serum creatinine ( Cr)≤1.5×ULN or calculate the creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula method.
11. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography.
12. Life expectancy ≥3 months.
13. Agree to use at least one medically approved contraceptive method during the trial period and at least 6 months after the last dose (female patients: such as intrauterine devices, contraceptives or condoms, etc.; male patients: such as condoms, abstinence, etc.). Female patients must be non-lactating.
14. Subjects must be fully informed of the content, process and possible risks and benefits of the research and sign the informed consent form. Good compliance, able to complete the study and follow-up.

Exclusion Criteria:

1. Known to have severe hypersensitivity to any monoclonal antibody (≥CTCAE grade 3).
2. Not recovered from the adverse reactions caused by previous anti-tumor treatments (≥CTCAE grade 1), excluding hair loss, pigmentation, and fatigue.
3. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
4. Received any live vaccines within 4 weeks before enrollment.
5. Have undergone surgery within 4 weeks before enrollment, and the investigator believes that the patient's state has not recovered to the point where the study can be started.
6. Have a history of hemolytic disease, immune-mediated thrombocytopenia, or Evans syndrome within 3 months before enrollment. Currently suffering from active or suspicious autoimmune disease or a history of autoimmune disease within the past 2 years.
7. Phase Ia and Ib: previous exposure to any CD47 antibody, SIRPα antibody or CD47/SIRPα recombinant protein, or previous exposure to any anti-programmed death receptor 1 (PD-1) or anti-programmed death ligand 1 ( PD-L1) antibody.
8. Received any systemic anti-tumor therapy within 4 weeks before enrollment.
9. Participated in other clinical trials within 4 weeks before enrollment and used clinical investigational drugs during this period.
10. Central nervous system metastases with clinical symptoms were found within 4 weeks before enrollment. Patients who have previously received treatment for brain or meningeal metastases, if clinical stability has been maintained for at least 2 months, and have stopped systemic hormone therapy (dose>10 mg/day prednisone or other curative hormones) for more than 4 weeks can be included.
11. Patients with ascites (ascites), pleural effusion (pleural effusion) or pericardial effusion that cannot be controlled by drainage or other methods.
12. Past or present suffering from other malignant tumors (except for cured skin basal cell carcinoma and cervical carcinoma in situ).
13. Suffering from serious or poorly controlled diseases, including but not limited to: ① Myocardial infarction, arrhythmia, congestive heart failure, etc. that require treatment or intervention occurred within 3 months before enrollment. ②Human immunodeficiency virus (HIV) infection (HIV antibody positive); hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive and HBV DNA ≥500 IU/mL or ≥1×10^3 copies/mL) ; HCV antibody positive and HCV RNA positive. ③ Poorly controlled diabetes, hypertension, thyroid disease, etc.; ④Severe and uncontrollable lung diseases (severe infectious pneumonia, interstitial lung disease, etc.) (≥CTCAE grade 3); ⑤Uncontrolled serious Infection (≥CTCAE grade 3).
14. With any situations that the researcher considers inappropriate to participate in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Dose limiting toxicities (DLTs) (Phase Ⅰ) | 28 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
Objective response rate (ORR) in dose expansion (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1 or Lugano 2014.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmax) following single dose.
Pharmacokinetic (PK) Tmax (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-t ) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) t1/2 (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,max) following single dose.
Pharmacokinetic (PK) Css,min (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,min) following single dose.
Pharmacokinetic (PK) AUCss (Phase Ⅰ) | Day1，2，3，7，14，21, 28 of DLT observation period , Day1of each subsequent cycle (each cycle is 7 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUCss) following single dose.
Objective response rate (ORR) in dose escalation (Phase Ⅰ) | Baseline through up to 2 years or until disease progression
  Tumor response based on RECIST 1.1 or Lugano 2014.
Incidence of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IBC0966 (Phase Ⅰ) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IBC0966.(Phase Ⅰ)
Progression free survival (PFS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1 or Lugano 2014.
Overall survival (OS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1 or Lugano 2014.
Disease control rate (DCR) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1 or Lugano 2014.
Incidence of adverse events (AEs) and SAEs (Phase Ⅱa) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IBC0966 (Phase Ⅱa) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IBC0966.(Phase Ⅱa)

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhang, Principal Investigator — The Affiliated Tumor Hospital of Harbin Medical University
Locations (1):
- The Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No